CLINICAL TRIAL: NCT06107335
Title: Effect of Albumin Versus Routine Care on Hemodynamic Response and Stability in Patients With Preeclampsia Guided by a Non-invasive Hemodynamic Monitoring System During Cesarean Delivery With Spinal Anesthesia - A Randomized Controlled Study
Brief Title: Effect of Albumin Versus Routine Care on Hemodynamic Response and Stability in Patients With Preeclampsia Guided by a Non-invasive Hemodynamic Monitoring System During Cesarean Delivery With Spinal Anesthesia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Onyi C Onuoha, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-23-0090
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Pre-Eclampsia
Keywords: Pre-Eclampsia; Albumin; Hemodynamic
MeSH Terms: conditions — Pre-Eclampsia | interventions — Serum Albumin, Human; Colloids; Albumins; Ringer's Lactate; Crystalloid Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fluid restriction using crystalloid (Active Comparator): Fluid restriction will be achieved with the crystalloid lactated ringer's injection administered at at a keep-the-vein-open (KVO) rate of 75 milliliters per hour (mL/hr).
  Interventions: Drug: Lactated Ringer's Injection (crystalloid)
- Fluid replacement using colloid as guided by stroke volume variation (SVV) (Experimental): Fluid replacement will be achieved with the colloid 5% albumin infusion. Use of colloid will be guided by stroke volume variation (SVV) as assessed by the Edwards HemoSphere monitor with ClearSight-Acumen finger cuff device.
  Interventions: Drug: Human Albumin (colloid); Device: Edwards HemoSphere monitor with ClearSight-Acumen finger cuff

INTERVENTIONS:
Drug: Human Albumin (colloid) — Fluid replacement will be achieved with colloid (5% albumin infusion). A bolus infusion of up to 500 milliliters (mL) of 5% Albumin will be administered prior to the placement of neuraxial anesthesia. If stroke volume variation (SVV) drops to less than 13% during the infusion of albumin, the infusion will be halted. At the completion of the placement of the spinal/combined spinal-epidural (CSE) anesthesia, study participants will receive the remaining albumin infusion if it was initially halted and SVV increases back to >13% during the procedure (to a total maximum of 500 mL albumin for the entire procedure).
  Other Names: Albutein
  Arms: Fluid replacement using colloid as guided by stroke volume variation (SVV)
Drug: Lactated Ringer's Injection (crystalloid) — Fluid restriction will be achieved with crystalloid (lactated ringer's injection) administered at a keep-the-vein-open (KVO) rate of 75 milliliters per hour (mL/hr), administered during the procedure.
  Arms: Fluid restriction using crystalloid
Device: Edwards HemoSphere monitor with ClearSight-Acumen finger cuff — Use of colloid will be guided by stroke volume variation (SVV) as assessed by the Edwards HemoSphere monitor with ClearSight-Acumen finger cuff device. The Edwards HemoSphere monitor with ClearSight-Acumen (CSA) finger cuff is a hemodynamic monitoring system that obtains continuous blood pressure readings from a cuff on the finger. In study participants, the finger cuff will be placed on the middle finger of one of the hands. The Edwards device can be used to predict impending intraoperative hypotension before its occurrence. The device has the ability to assess vasodilatory status using systemic vascular resistance (SVR), volume status using stroke volume variation (SVV) and stroke volume (SV) and the use of Carbon Monoxide (CO) to assess for underlying cardiac suppression. It also incorporates the hypotension prediction index (HPI), an algorithm that uses the arterial waveform to predict early phases of intraoperative hypotension.
  Arms: Fluid replacement using colloid as guided by stroke volume variation (SVV)

SUMMARY:
The purpose of this study is to compare the effect of albumin versus routine care on hemodynamic response and stability in pre-eclamptic patients during cesarean delivery. The hypothesis is that volume replacement with albumin guided by stroke volume variation (SVV) using a ClearSight-Acumen (CS-A) monitor, before cesarean delivery (CD), improves hemodynamic stability in preeclamptic patients with severe features compared to routine care, under neuraxial anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age greater or equal to 24 weeks
* Diagnosis of preeclampsia with severe features [Pre-eclampsia is defined as high blood pressure after 20 weeks with or without proteinuria. Pre-eclampsia with severe features is defined as the presence of preeclampsia with any of the following features: severe hypertension (blood pressure ≥160/110 mmHg on two separate occasions); thrombocytopenia (platelet count <100,000 per microliter); impaired liver function (elevated liver transaminases to twice the normal concentration or severe persistent right upper quadrant or epigastric pain not responsive to medications); progressive renal insufficiency with a serum creatinine level of >1.1 mg/dl or doubling of the serum creatinine level in the absence of other renal disease; pulmonary edema or unexplained new-onset cerebral symptoms (headache) unresponsive to medications or visual disturbances.]
* Scheduled Cesarean Delivery
* Unscheduled Cesarean Delivery with the goal to proceed to the operating room within no less than 30 minutes due to concern for maternal or fetal status that is not immediately life threatening.
* Requiring Neuraxial Anesthesia (spinal or CSE)

Exclusion Criteria:

* Patient declines to participate in the study
* Labor
* Contraindications to the use of neuraxial anesthesia (coagulopathy, infection at the insertion site, intracranial mass etc.)
* Unscheduled Cesarean Delivery with the goal to proceed to the operating room immediately for delivery of the baby due to imminent/unavoidable threat to the life of the mother or fetus.
* The use of or conversion to General Anesthesia
* Non-reassuring fetal status including the presence of cardiac or multi-system anomalies, category III tracing etc.
* Significant maternal cardiopulmonary disease including pulmonary hypertension, ischemic heart disease with systolic dysfunction, pulmonary edema etc.
* Significant intraoperative events (such as hemorrhage) requiring administration of multiple blood products and ICU admission.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with fluid responsiveness | from baseline to thirty minutes after arrival to the Post Anesthesia Care Unit (PACU)
  "Fluid responsiveness" (in other words, a "positive response") is defined as a volume-induced correction to stroke volume variation (SVV) values < 13%. SVV measurements will be made using the Edwards HemoSphere monitor with ClearSight-Acumen finger cuff.

SECONDARY OUTCOMES:
Number of participants with fluid responsiveness stability | from baseline to thirty minutes after arrival to the Post Anesthesia Care Unit (PACU)
Maternal blood pressure (diastolic) | baseline, after infusion of study intervention, at completion of placement of the spinal/CSE anesthesia, at completion of delivery of the baby, at end of procedure when leave operating room, thirty minutes after arrival to PACU
Maternal blood pressure (systolic) | baseline, after infusion of study intervention, at completion of placement of the spinal/CSE anesthesia, at completion of delivery of the baby, at end of procedure when leave operating room, thirty minutes after arrival to PACU
Total amount in milligrams of rescue vasopressor drug given | from start of operation to thirty minutes after arrival to the Post Anesthesia Care Unit (PACU)
Number of adverse events | from start of operation to discharge from the Post Anesthesia Care Unit (PACU)

CONTACTS AND LOCATIONS:
Overall Officials: Onyi Onuoha, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No